CLINICAL TRIAL: NCT03967886
Title: A Randomized, Double-blind, Placebo-controlled, Multi-centers Clinical Trial to Assess the Efficacy and Safety of YYD601 in NERD Patients (Phase3).
Brief Title: Clinical Trial to Assess the Efficacy and Safety of YYD601 in NERD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YYPCT_YYD601_P3(2)
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YYD601 20mg (Experimental): Esomeprazole magnesium Dihydrate.
  Interventions: Drug: YYD601 20mg; Drug: Placebos
- Nexium 20mg (Active Comparator): Esomeprazole magnesium trihydrate, a substituted benzimidazole.
  Interventions: Drug: Nexium 20mg; Drug: Placebos

INTERVENTIONS:
Drug: YYD601 20mg — Patients should take drugs an hour before breakfast.
  Arms: YYD601 20mg
Drug: Nexium 20mg — Patients should take drugs an hour before breakfast.
  Arms: Nexium 20mg
Drug: Placebos — The placebo YYD601 is made from microcrystalline cellulose covered with hard shell. The placebo Nexium is made from microcrystalline cellulose, Crospovidone, Magnesiumstearat and other ingredients.

SUMMARY:
Clinical Trial to Assess the Efficacy and Safety of YYD601 in NERD Patients

DETAILED DESCRIPTION:
This Phase 3 Clinical Trial is Designed as Randomized, Double-blind, Placebo-controlled, Multi-centers Clinical Trial to Assess the Efficacy and Safety of YYD601 in NERD Patients (Phase3).

ELIGIBILITY:
Inclusion Criteria:

* A man or woman over 20 years old less than 70 years old.
* A man or woman who has below all characters and diagnosis as NERD.

  1. A man or woman who has experienced symptom(hearburn or/and acid regurgitation) over 3month at least.
  2. A man or woman who has experienced symptom(heartburn or/and acid regurgitation) within 7days before Visit1, meet below 1) or 2) criteria.

     ** Symptom (heartburn and acid regurgitation) is confirmed by RDQ
     * Experienced above 2 days in a week, heartburn of acid regurgitation above the weakness.
     * Experienced above 1 day in a week, heartburn of acid regurgitation above the middle.
  3. A man or woman who has been made diagnosis as LA grade0(Zero) measured through the dendoscopy which is corried out within 14 days, there is no observed muscosal break.
* A man or woman who has a full understanding of this clinical trial through the detailed explanation, agree in writing to participate in this trial.

Exclusion Criteria:

* Who has hyper sensitivity reaction about other drugs, ingredients, components of investigator product or compound of benzimidazole.
* Who has ERD.
* Who get a diagnosis as a IBS within the last 3 months.
* Who have taken drugs about reflux esophagitis (H₂-receptor inhibitor (H2RA) Prostaglandin(PG), Antacid, Prokinetic acid etc.) above 2 times as an usual dose. (* refer to the Concomitant medication in text.)
* Who havbe taken gastric acid secretion inhibitors including PPIs within 2 weeks before the endoscopy.
* Who has been experienced the disease affecting the esophagus(Eosinophilic esophagitis, esophageal varices, cirrhosis, Virus or Fungal infection, Esophageal stricture, primary esophageal motility disorder and gastrointestinal bleeding). Or who has a history of radio therapeutics, freeze treatment about the esophagus.
* Who has the gastric or duodenal ulcer, Zollinger-Ellison and other acid hypersecretory condition been experienced.
* Who has hyper-sensitivity, reaction about PPIs (ex. Lansoprazole, omeprazole, rabeprazole, pantoprazole or esomeprazole).
* Who has gotten a diagnosis as a cancer within 5 years before participated in this clinical trail (expect the basal cell on the skin), peptic ulcer or benign tumor.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Recovered percentage(%) of the symptom | within 4 weeks
  Recovered percentage(%) of the symptom(heartburn or/and acid regurgitation) measured by RDQ after administration(baseline).
Change of the score about the symptom | within 4 weeks
  Change of the score about the symptom(heartburn or/and acid regurgitation) measured by RDQ after administration(baseline).
Percentage(%) of the patients who have symptom during the daytime | within 4 weeks
  Percentage(%) of the patients who have symptom(heartburn or/and acid regurgitation) during the daytime measured by Patients diary after administration(baseline).
Percentage(%) of the patients who have symptom during the nighttime | within 4 weeks
  Percentage(%) of the patients who have symptom(heartburn or/and acid regurgitation) during the nighttime measured by Patients diary after administration(baseline).
Percentage(%) of the days no symtom | within 4 weeks
  Percentage(%) of the days no symptom(heartburn or/and acid regurgitation) among the patients who have symptom(heartburn or/and acid regurgitation) during the nighttime measured by Patients diary after administration(baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Seoul, South Korea